CLINICAL TRIAL: NCT04049110
Title: SGLT-2 Inhibition Using Dapagliflozin During and After Physical Exercise - Effects on Glycemic Variability, Hormonal Regulators of Glucose Homeostasis and Ketone Body in Type 1 Diabetes - a Randomized, Placebo-controlled, Open-label, Cross-over Intervention Study
Brief Title: Dapagliflozin in Physical Exercise in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CUI_002_02
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, open-label, crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin first, placebo second (Experimental): Dapagliflozin followed by placebo
  Interventions: Drug: Forxiga 10mg; Drug: Placebo
- Placebo first, Dapagliflozin second (Experimental): Placebo followed by dapagliflozin
  Interventions: Drug: Forxiga 10mg; Drug: Placebo

INTERVENTIONS:
Drug: Forxiga 10mg — Dapagliflozin 10mg per 24 hours, oral, for 7 consecutive days
  Other Names: Dapagliflozin
Drug: Placebo — Placebo 1 tablet per 24 hours, oral, for 7 consecutive days

SUMMARY:
Inhibitors of sodium-dependent glucose-transporter 2 (SGLT-2 inhibitors, including dapagliflozin) inhibit glucose reabsorption in renal tubular cells, hereby increasing glycosuria in the hyperglycemic state. Its mechanisms of action are independent of insulin, which makes SGLT-2 inhibitors a potential adjunct to insulin in type 1 diabetes mellitus (T1DM).

However, a higher risk for diabetic ketoacidosis (DKA) was reported in patients with T1DM taking SGLT-2 inhibitors. DKA depends on an accumulation of ketone bodies in the blood stream, which equals an accumulation of acids that lead to acidosis. The underlying mechanisms of this observation are unknown. Ketone body production depends on the molar ratio of glucagon to insulin, with insulin suppressing but glucagon stimulating ketone body production. This translates into higher production during relative insulin deficiency, carbohydrate deficiency, and prolonged fasting, which occurs during sickness but also physical exercise. Physical exercise is a recommended cornerstone in the treatment of T1DM and current treatment guidelines recommend both, reductions of insulin doses and ingestion of additional carbohydrates to avoid hypoglycemic events. These adaptions might increase relative insulin deficiency, hyperglycemia and glycaemic variability, which might in turn promote ketone body production. The addition of SGLT-2 inhibitors further may promote ketogenesis even though there are reports of SGLT-2 inhibitors increase Glucagon-like-peptide-1 (GLP-1) in patients with T1DM. GLP-1 is a suppressor of glucagon secretion. In summary, knowledge about the effects of SGLT-2 inhibition on ketone body production is scarce, especially during exercise in patients with T1DM.

The study seeks to illustrate the effect of SGLT-2 inhibition on glycemic variability and ketone body production during and after recreational exercise in patients with T1DM. The results of study 2 will provide the basis for future studies investigating the underlying mechanisms of potentially modified ketone body production during and after exercise under SGLT-2 inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosis of T1DM
* Duration of T1DM > 5 years
* Male or female sex
* Insulin therapy via multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII)
* Body mass index (BMI) between 20 and 29 kg/m2
* Adherence to sufficient contraceptive measures (double barrier method combining hormonal with mechanical barriers).
* Ability to perform a 60 minutes exercise session at 50% VO2max.

Exclusion Criteria:

* Diagnosis of renal and/or hepatic dysfunction
* History of malignancy of any kind
* Intake of drugs influencing glucose homeostasis during the last three months
* Alcohol or drug abuse
* Inadequate vein status on both forearms
* Active smoker
* Known pregnancy, positive plasma beta human choriogonadotropine test prior to study inclusion or intention to become pregnant during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Mean Amplitude of Glucose Excursions (MAGE) after physical exercise | From completion of physical exercise at day 7 of each intervention period to 72 hours after
  MAGE will be calculated via sensor glucose measurements obtained over 72 hours after physical exercise

SECONDARY OUTCOMES:
Area under the curve for glucagon-like peptide I before, during and after physical exercise | From time-point 0 to 120 minutes before, during and after physical exercise session
  Glucagon-like peptide I will be measured at the beginning, during and after physical exercise following each intervention period
Area under the curve for glucagon before, during and after physical exercise | From time-point 0 to 120 minutes before, during and after physical exercise session
  Glucagon will be measured at the beginning, during and after physical exercise following each intervention period

OTHER OUTCOMES:
Area under the curve for ketone bodies before, during and after physical exercise | From time-point 0 to 120 minutes before, during and after physical exercise session
  Ketone bodies will be measured at the beginning, during and after physical exercise
Area under the curve for free fatty acids bodies before, during and after physical exercise | From time-point 0 to 120 minutes before, during and after physical exercise session
  Free fatty acids will be measured at the beginning, during and after physical exercise
Area under the curve for somatostatin before, during and after physical exercise | From time-point 0 to 120 minutes before, during and after physical exercise session
  Somatostatin will be measured at the beginning, during and after physical exercise

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, Prof. MD, Principal Investigator — Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, University Clinics Bern, Inselspital, Bern, Switzerland
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: From July, 30th 2021 ongoing
Access Criteria: Contact with the Study Sponsor